CLINICAL TRIAL: NCT00424983
Title: A Stratified, Randomized, Open-label, Multi-center Comparative 2-arm Trial of PK, PD, and Safety of Zoledronic Acid Infusions Administered Monthly vs. Every 3-month, in Multiple Myeloma Patients With Malignant Bone Lesions, and Breast Cancer Patients With Bone Metastasis, Who Have Received 9-12* Doses of Zoledronic Acid Over the Prior Year. (*Amendment 1 Changed the Required Doses to 9-20 But Due to FDA Guidelines, the Title Has Not Been Changed)
Brief Title: Study of Zoledronic Acid Administered Monthly Versus Every 3 Months in Multiple Myeloma and Breast Cancer Patients Who Were Treated With Zoledronic Acid the Prior Year
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446E2105; 2007-004719-73 (EudraCT Number)
Record Dates: First submitted 2007-01-19; First posted 2007-01-22 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2014-09

CONDITIONS: Multiple Myeloma; Breast Cancer
Keywords: Multiple myeloma; breast cancer; zoledronic acid; pharmacokinetics
MeSH Terms: conditions — Multiple Myeloma; Breast Neoplasms | interventions — Zoledronic Acid

ARMS (2):
- Zometa q 4 weeks (Experimental)
  Interventions: Drug: Zoledronic acid
- Zometa q 12 weeks (Active Comparator)
  Interventions: Drug: Zoledronic acid

INTERVENTIONS:
Drug: Zoledronic acid
  Other Names: ZOL446

SUMMARY:
The primary objective of this study is to investigate the repeat-dose pharmacokinetic (PK) profile of zoledronic acid when administered every 4 weeks versus every 12 weeks, in patients treated with 9-20 infusions of zoledronic acid during the previous 10-15 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18-75 years of age
* Multiple myeloma or breast cancer with bone involvement
* Treatment with zoledronic acid for bone lesions between 10-15 months prior to entry into study with a total of 9-20 infusions received.

Exclusion Criteria:

* Current active dental problems or recent (within 8 weeks) or planned dental or jaw surgery
* Active or uncontrolled infection, liver, or renal disease
* History of treatment with intravenous bisphosphonates
* Diagnosis of metabolic bone disorders other than osteoporosis (e.g. Paget's disease)

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-11; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Sequential plasmas concentrations of zoledronic acid collected at 13 study visits between visit 2 to visit 17 | every four (4) weeks
Sequential urine concentrations of zoledronic acid collected at 9 study visits between visit 2 to visit 13 | every four (4) weeks

SECONDARY OUTCOMES:
Pharmacodynamic outcomes will be measured by the concentration of bone resorption markers at all visits. | every four (4) weeks
Efficacy outcomes will be measured throughout the study by number and time to skeletal related events (determined by bone surveys and bone scans) as well as the measurement of pain and analgesic scores. | bone survey = every 12 weeks; bone scan = every 24 weeks; pain & analgesic scores = weekly prior to visit 8 (inclusive), every 4 weeks after visit 8

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis, Study Chair — Novartis
Locations (7):
- United States (7):
  - Oncotherapeutics, West Hollywood, California
  - Rocky Mountain Cancer Centers RMCC, Greenwood Village, Colorado
  - Norwalk Hospital, Norwalk, Connecticut
  - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Huntsman Cancer Institute Univ. of Utah, Salt Lake City, Utah
  - University of Vermont Fletcher Allen Health Care, Burlington, Vermont
  - Virginia Cancer Institute Virginia Cancer Center, Richmond, Virginia

REFERENCES:
- See also: Visit NovartisClinicalTrials.com: Pre-qualify for a trial, and view a list of trials and participating study centers. — https://www.novartisclinicaltrials.com/TrialConnectWeb/home.nov
- See also: Results for CZOL446E2105 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=7464